CLINICAL TRIAL: NCT01301443
Title: A Phase I Dose Escalation Safety Study of Subretinally Injected RetinoStat, a Lentiviral Vector Expressing Endostatin and Angiostatin, in Patients With Advanced Neovascular Age-Related Macular Degeneration
Brief Title: Phase I Dose Escalation Safety Study of RetinoStat in Advanced Age-Related Macular Degeneration (AMD)
Acronym: GEM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS1/001/10
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Subretinally Injected RetinoStat (Experimental): Subretinally injected RetinoStat
  Interventions: Drug: Subretinally injected RetinoStat

INTERVENTIONS:
Drug: Subretinally injected RetinoStat — Single subretinal injections, with increasing doses. 9 patients with 3 patients at each dose followed, by 12 patients at maximum tolerated dose.
  Other Names: OXB-201

SUMMARY:
The purpose of this first in man study is to examine the safety of an experimental gene transfer agent, RetinoStat, designed to treat neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
There are two parts to the study. A dose-escalation phase looking at three doses of RetinoStat starting with the lowest dose, three patients will be recruited at each dose level. The escalation phase will be followed by a dose confirmation phase where the highest dose that is safe and well tolerated will be examined in 9 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AMD with active CNV that shows evidence of leakage.
* BCVA less than or equal to 20/200 in the study eye for dose escalation phase.
* BCVA less than or equal to 20/80 in the study eye for maximum tolerated dose phase.

Exclusion Criteria:

* Significant ocular abnormalities that prevent retinal assessment.
* Treatment with steroids within three months of screening.
* Treatment with anti-VEGF therapy to either eye within one month of screening.
* Clinically significant intercurrent illnesses, laboratory, ECG or chest XRay abnormalities.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events | 24 weeks
  The number and percentage of patients with treatment emergent adverse events.

SECONDARY OUTCOMES:
Change from baseline in subretinal and intraretinal fluid as measured by OCT | 24 weeks
  The change from baseline in the amount of subretinal and intraretinal fluid measured by Optical Coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University Hospital
Locations (3):
- United States (3):
  - The University of Iowa, Iowa City, Iowa
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Dr Andreas Lauer - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Campochiaro PA, Lauer AK, Sohn EH, Mir TA, Naylor S, Anderton MC, Kelleher M, Harrop R, Ellis S, Mitrophanous KA. Lentiviral Vector Gene Transfer of Endostatin/Angiostatin for Macular Degeneration (GEM) Study. Hum Gene Ther. 2017 Jan;28(1):99-111. doi: 10.1089/hum.2016.117. Epub 2016 Sep 26. PMID 27710144